CLINICAL TRIAL: NCT00347347
Title: Comparative Study of Cycloplegic Refraction and Subjective Refraction With Fogging in School Age Children
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other)
Other Study IDs: R456/05/2006
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-05

CONDITIONS: Myopia; Refractive Error
MeSH Terms: conditions — Myopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
A thorough ophthalmic examination of a child must include a refraction and this is often done with cycloplegia. In our study, we aim to determine at which age group a non-cycloplegic refraction technique closely correlates with a cycloplegic refraction and hence, would obviate the need for cycloplegic refraction in our routine clinical practice.

DETAILED DESCRIPTION:
The accommodative response in young phakic patients has been known to result in over-estimation of myopia and subsequently inappropriate prescriptions. Therefore, the rationale for cycloplegia is to inhibit the accommodative response in order to obtain a true measurement of the refractive error.

Different cycloplegic agents have been in common use for the last five decades. Cyclopentolate is widely used and is commercially available in concentrations of 0.5% and 1%. Tropicamide is another widely used cycloplegic agent and is available in 0.5% and 1% concentrations.

The advantages of a non-cycloplegic technique would be firstly, the avoidance of any possible harmful effects from the cycloplegic agents used. Secondly, it would vastly reduce waiting times for parents and children and allow for a much more efficient clinical service. Finally, there may be a significant cost-saving feature involved if these cycloplegic agents are no longer required.

This will be a prospective clinical audit/survey involving children between the ages of 4 years and 13 years who attend the paediatric ophthalmology clinics in KK Women's and Children's Hospital as well as the Singapore National Eye Centre.

All eligible children will have had a cycloplegic refraction and a non-cycloplegic refraction with fogging. A survey of children between the ages of 4 and 13 years who have had refraction with both these techniques will be undertaken and the difference in spherical error between the 2 techniques will be recorded for each child. We aim to accumulate 15 children from each age group.

ELIGIBILITY:
Inclusion Criteria:

1. As part of the ophthalmic evaluation, will undergo non-cycloplegic and cycloplegic refraction.
2. Informed consent has been obtained from a parent or guardian.
3. Aged between 4 years and 13 years old.
4. Able to cooperate with examination(s) as stated.

Exclusion Criteria:

1. Known allergy or adverse reaction to cyclopentolate.
2. Unable to cooperate with examination(s) stated.
3. Parent or guardian objection.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 4-13 years old.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Mean spherical error (MSE) of less than or equal to 0.50D between the non-cycloplegic and cycloplegic refractive results .
MSE calculated by subtracting the non-cycloplegic spherical error from the cycloplegic spherical error.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Ling, FRCS(G), Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore